CLINICAL TRIAL: NCT06835556
Title: Testing the Role of Belief Updating in Persecutory Delusions
Brief Title: Volatility in Paranoia (VIP) Trial: An RCT of Changes in Volatility With Psychotherapy
Acronym: VIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Julia Sheffield, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 240788; R01MH137024 (NIH)
Record Dates: First submitted 2025-02-12; First posted 2025-02-19 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia Disorders
Keywords: Schizophrenia; Delusion; Paranoia; Psychotherapy; Beliefs; Volatility; Cognitive Behavioral Therapy; CBTp; Psychosis
MeSH Terms: conditions — Schizophrenia; Delusions; Paranoid Disorders; Psychotic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBTp (Experimental): Weekly individual psychotherapy targeting specific maintenance factors of paranoia (worry, anomalous experiences, self-confidence, and safety behaviors), tailored to the participant's experience
  Interventions: Behavioral: Cognitive Behavioral Therapy
- TAU + Phone Check-In (Active Comparator): Participants will continue with their regular care (treatment as usual (TAU)) without interference from the study team. In addition to TAU, a study therapist will call them weekly to review what treatment the participants have engaged in. Phone calls will last approximately 5-10 minutes
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Individuals will be assessed for which psychological factors are maintaining paranoia in their daily lives. They will collaboratively identify one maintenance factor to focus on (e.g. worry, anomalous experience, self-confidence, PTSD) for 8 weeks of individual therapy. Then, all participants will transition to 8 weeks of individual therapy focused on dropping safety behaviors and re-engaging in everyday life.
  Arms: CBTp
Behavioral: TAU — Individuals will continue treatment as usual (TAU). In addition they will have contact with a study therapist weekly via phone to provide information on what treatment they received. Phone check-ins will last approximately 5-10 minutes.
  Arms: TAU + Phone Check-In

SUMMARY:
The goal of this clinical trial is to learn whether learning and belief updating change in response to the treatment of persecutory delusions, in individuals with schizophrenia-spectrum disorders.

The main questions are:

1. do prior expectations about environmental volatility reduce following effective psychotherapeutic treatment of delusions?
2. does corresponding brain activity related to volatility change with effective treatment of delusions?

Participants will:

1. engage in CBTp or TAU + phone check-ins for 16 weeks
2. complete assessments at 4 timepoints over the course of 6 months
3. complete an MRI when possible

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 - 65.
* Communicative in English.
* Premorbid IQ >79 (WTAR)
* Provide voluntary, written informed consent.
* Stable medication regimen over at least the past two weeks, including the use of either an oral or intramuscular administration of an antipsychotic medication.
* Diagnosis of a non-affective psychotic disorder (e.g. schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder)
* A persecutory delusion scoring at least a 3 on the conviction scale of the Psychotic Symptoms Rating Scale (PSYRATS) that had persisted for at least two months and that was not considered the direct result of substance use.

Exclusion Criteria:

* Serious medical or neurological illness known to interfere with cognitive functioning (uncontrolled/unstable diabetes, uncontrolled hypothyroidism, Cushing's disease, Lupus, any demyelinating disease such as Multiple Sclerosis, HIV infection, CNS infection, unstable heart disease, active hepatitis, other significant endocrine condition, any cancer involving the CNS/brain, any uncorrected vision problems, tardive dyskinesia).
* History of severe head trauma with loss of consciousness >30 minutes.
* Primary diagnosis of alcohol or substance use disorder or personality disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2029-09-03 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in prior expectations of volatility (mu3) | Baseline to 16 weeks
  Reversal learning data will be collected from a 3-option probabilistic reversal learning task. This data will be analyzed using a computational model that estimates the prior expectations of environmental volatility. That parameter, in many models, is Mu3.
Change in unexpected uncertainty (kappa) | Baseline to 16 weeks
  Reversal learning data will be collected from a 3-option probabilistic reversal learning task. This data will be analyzed using a computational model that estimates the unexpected uncertainty, sometimes also referred to as sensitivity to volatility.
Change in psychotic Symptom Rating Scale (PSYRATS)- Belief Subscale Total | Baseline to 16 weeks
  The PSYRATS is a interview-assisted assessment measuring the severity of a delusional belief. Total scores range from 0-24 with high scores indicating more severe delusion; 6 questions, 0-4 scale for each item
Change in PANSS Positive Symptoms - Total | Baseline to 16 weeks
  The PANSS is a 30-item clinician-rated instrument for assessing schizophrenia symptoms. It consists of 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score for each participant was sum of the rating assigned to each of the 30 PANSS items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. The positive symptom total score is the sum of the Positive Symptom items
BOLD activation change during PRL task, pre/post treatment - prefrontal cortex | Baseline to 16 weeks
  functional MRI will be used to collect BOLD activation data during the PRL reversal learning task. The investigators expect changes in activation following treatment, particularly in the CBTp group
BOLD activation change pre/post treatment - striatum | Baseline to 16 weeks
  functional MRI will be used to collect BOLD activation data during the PRL reversal learning task. The investigators expect changes in activation following treatment, particularly in the CBTp group
BOLD activation change during PRL task, pre/post treatment - locus coeruleus | Baseline to 16 weeks
  functional MRI will be used to collect BOLD activation data during the PRL reversal learning task. The investigators expect changes in activation following treatment, particularly in the CBTp group
Task-based functional connectivity changes during PRL task, pre/post treatment - prefrontal cortex to striatum | Baseline to 16 weeks
  Functional connectivity during the PRL task will be quantified between the dlPFC and striatum

SECONDARY OUTCOMES:
Change in PANSS P1 Item | Baseline to 16 weeks
  The PANSS is a 30-item clinician-rated instrument for assessing schizophrenia symptoms. It consists of 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score for each participant was sum of the rating assigned to each of the 30 PANSS items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. P1 is the first item on the scale, representing delusion severity
Change in PANSS P6 Item | Baseline to 16 weeks
  The PANSS is a 30-item clinician-rated instrument for assessing schizophrenia symptoms. It consists of 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score for each participant was sum of the rating assigned to each of the 30 PANSS items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. P6 is the item on the scale assessing severity of paranoia/suspiciousness
Change in meta-volatility learning rate (omega3) | Baseline to 16 weeks
  Reversal learning data will be collected from a 3-option probabilistic reversal learning task. This data will be analyzed using a computational model that estimates the meta-volatility.
BOLD activation changes during PRL task, pre/post treatment - whole brain analysis | Baseline to 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP